CLINICAL TRIAL: NCT02225964
Title: Multi-modality MRI Study on Differences in Conversion of aMCI Patients With APOEε4 to AD
Status: Completed | Type: Observational
Sponsor: XuanwuH 2 (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Chief physician, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: XuanwuH 2
Record Dates: First submitted 2014-08-24; First posted 2014-08-26 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Mild Cognitive Impairment
Keywords: APOEε4
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aMCIp,aMCIs: progressive aMCI,stable aMCI

SUMMARY:
This study is to find out the imaging marker and the changing laws of the marker during the course of the disease. The final purpose is to provide scientific evidence for new prevention, diagnosis and treatment of Alzheimer's disease.

DETAILED DESCRIPTION:
It is an urgent problem in the field of cognitive neuroscience to tell the conversion progression of amnestic mild cognitive impairment(aMCI) patients with Apolipoproteinε4(APOEε4) to Alzheimer's Disease(AD). Based on our preliminary work, we will study the special group of aMCI patients with APOEε4 with multi-modality magnetic resonance imaging (resting-state functional MRI, structural MRI and diffusion tensor imaging) longitudinally. Besides, we will also detect the APOE genotype of each sample and enlarge the sample size. According to situation of the conversion or non-conversion and differences in the conversion progression, we will analyze the data between the inter-groups and intra-groups, compare the imaging data of baseline and follow-up, find the prediction imaging marker of AD and optimize the reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

* Complaint about memory loss and confirmed by an informant
* Cognitive impairment in single or multiple domains, adjusted for age and education
* Normal or near-normal performance on general cognitive function and no or minimum impairment of daily life activities
* A Clinical Dementia Rating (CDR) score is 0.5
* Failure to meet the criteria for dementia
* Carrying susceptible gene APOEε4
* Must be able to accept examination of MRI, sight and hearing allow to complete test

Exclusion Criteria:

* Other diseases that cause cognitive impairment,such as thyroid disease,stroke and so on
* people who have severe visual and hearing impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: aMCI patients with APOEε4
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
the conversion of aMCI patients with APOEε4 to AD | one year
  According to situation of the conversion or non-conversion and differences in the conversion progression, we will analyze the data between the inter-groups and intra-groups, compare the imaging data of baseline and follow-up, find the prediction imaging marker of AD and optimize the reliability and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurolgy,Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin H, Li M, Zhan Y, Lin L, Yang K, Hu S, Han Y. Disrupted white matter functional connectivity in aMCI APOEepsilon4 carriers: a resting-state study. Brain Imaging Behav. 2021 Aug;15(4):1739-1747. doi: 10.1007/s11682-020-00367-7. PMID 32715396
- [Derived] Yang L, Yan Y, Wang Y, Hu X, Lu J, Chan P, Yan T, Han Y. Gradual Disturbances of the Amplitude of Low-Frequency Fluctuations (ALFF) and Fractional ALFF in Alzheimer Spectrum. Front Neurosci. 2018 Dec 20;12:975. doi: 10.3389/fnins.2018.00975. eCollection 2018. PMID 30618593
- [Derived] Chen GQ, Sheng C, Li YX, Yu Y, Wang XN, Sun Y, Li HY, Li XY, Xie YY, Han Y. Neuroimaging basis in the conversion of aMCI patients with APOE-epsilon4 to AD: study protocol of a prospective diagnostic trial. BMC Neurol. 2016 May 12;16:64. doi: 10.1186/s12883-016-0587-2. PMID 27176479